CLINICAL TRIAL: NCT03125967
Title: Effects of Colored Light Exposure on Sleep Disturbance, Fatigue, and Functional Outcomes Following Acute Brain Injury
Brief Title: Daily Light Exposure for Sleep Disturbance, Fatigue, and Functional Outcomes in Acute Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Rehabilitation Institute (Other)
Collaborators: Washington State University (Other)
Responsible Party: Principal Investigator, Douglas L. Weeks, Director of Research, St. Luke's Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StLukesRI
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Traumatic Brain Injury; Non-traumatic Brain Injury
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: two-arm randomized placebo-controlled study with pre-exposure and post-exposure assessments
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue Light (Active Comparator): Blue light exposure (Philips GoLite Blu HF3429/60) administered daily for 25 minutes between 8:00AM and 9:00AM
  Interventions: Other: Philips GoLite Blu HF3429/60
- Red Light (Placebo Comparator): Red light exposure (Philips LivingColor Aura 70998/60/48) administered daily for 25 minutes between 8:00AM and 9:00AM
  Interventions: Other: Philips LivingColor Aura 70998/60/48

INTERVENTIONS:
Other: Philips GoLite Blu HF3429/60 — Exposure to daily morning colored light in the 440-485 nm wavelength range
  Arms: Blue Light
Other: Philips LivingColor Aura 70998/60/48 — Exposure to daily morning colored light in the 625-740 nm wavelength range
  Arms: Red Light

SUMMARY:
The purpose of this study is to assess the safety and efficacy of daily morning exposure to colored light in patients receiving acute inpatient rehabilitation services for stroke, traumatic brain injury, or non-traumatic brain injury with sleep disturbances such as poor nighttime sleep and/or excessive daytime sleepiness.In a two-arm randomized placebo-controlled study with pre-exposure and post-exposure assessments, we are comparing the effects of daily morning exposure to either blue light or red light on objective sleep quality, subjective sleep quality, functional rehabilitation outcomes, cognitive symptoms, fatigue, and neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient admission to St. Luke's Rehabilitation Institute for stroke, traumatic brain injury, or non-traumatic brain injury
2. Male or female, 18 to 85 years of age (to match limits of assessment instruments)
3. Able to provide written informed consent or have a legally authorized representative that can provide written informed consent
4. Stable neurologic status, as determined from subject's medical records and the study physician's opinion based on no new or changing symptoms
5. Normal vision or corrected to normal vision (if glasses or contacts are tinted, willing to remove during light exposure)
6. Normal hearing or corrected to normal hearing
7. Willing to complete baseline evaluations prior to inclusion in the study to include: sleepiness inventories, neuropsychological testing, self-report fatigue assessment

Exclusion Criteria:

1. History of epileptic or other seizure disorder
2. Cataract surgery in the past 12 months
3. Significant visual impairment affecting light reaching the retina/performance of the retina: cataracts, macular degeneration, diabetic retinopathy, congenital blindness, total blindness, glaucoma, or retinal detachment
4. Endorsement of suicidal ideation on the PHQ-9 depression screen (standard of care admission assessment at St. Luke's)
5. Pre-injury diagnosis of a sleep disorder, including: sleep apnea, insomnia, narcolepsy or periodic limb movement syndrome
6. Neurological disorders other than those attributed to the primary diagnosis, including multiple sclerosis, Parkinson's disease, Huntington's disease, Alzheimer's disease or other dementias, amyotrophic lateral sclerosis)
7. Bipolar diagnosis
8. Females who are pregnant as determined from subject's medical records or who are breastfeeding
9. In active withdrawal from alcohol or street drugs
10. Unwillingness to refrain from wearing tinted glasses or contact lenses during light exposure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time | From day of consent through study completion at discharge from inpatient rehabilitation, assessed for at least 10 days
  24/7 recording of total amount of time asleep via wrist-worn actigraph
Sleep Efficiency | From day of consent through study completion at discharge from inpatient rehabilitation, assessed for at least 10 days
  Recording of the proportion of time asleep relative to time in bed via wrist-worn actigraph
Sleep Fragmentation Index | From day of consent through study completion at discharge from inpatient rehabilitation, assessed for at least 10 days
  Recording of restlessness during a sleep period via wrist-worn actigraph
Frequency of Daytime Naps | From day of consent through study completion at discharge from inpatient rehabilitation, assessed for at least 10 days
  Recording of number of naps during daytime via wrist-worn actigraph

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale | Baseline and every 3 days plus at study completion, at least 10 days after consent
  Patient-report measure of daytime sleepiness
Wits Pictorial Sleepiness Scale | Baseline and every 3 days plus at study completion, at least 10 days after consent
  Patient-report measure of daytime sleepiness
Fatigue Visual Analog Scale | Baseline and every 3 days plus at study completion, at least 10 days after consent
  Patient-report measure of global fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Weeks, PhD, Principal Investigator — St. Luke's Rehabilitation Institute
Locations (1):
- St. Luke's Rehabilitation Institute, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weeks DL, Crooks E, O'Brien KE, Sprint G, Carter GT, Honn KA. A parallel-group randomized controlled trial of blue light versus red light for improving sleep, fatigue, and cognition following stroke: Pilot results and recommendations for further study. Contemp Clin Trials. 2024 Dec;147:107736. doi: 10.1016/j.cct.2024.107736. Epub 2024 Nov 6. PMID 39510247